CLINICAL TRIAL: NCT02583828
Title: Study in Letrozole Combined With Metronomic Oral Cyclophosphamide in Elderly Metastasis Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jun Ren MD, PhD, MD, PhD, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LET+CTX
Record Dates: First submitted 2015-10-13; First posted 2015-10-22 (Estimated); Last update posted 2024-02-07 (Actual); Status verified 2024-02

CONDITIONS: Breast Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Cyclophosphamide; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cyclophosphamide alone (Active Comparator): Patients who were resistant to letrozole will be randomized to receive cyclophosphamide alone or letrozole plus cyclophosphamide. Patients in this arm will receive cyclophosphamide 50 mg daily.
  Interventions: Drug: Cyclophosphamide 50mg
- Cyclophosphamide plus letrozole for resistant patients (Experimental): Patients who were resistant to letrozole will be randomized to receive cyclophosphamide alone or letrozole plus cyclophosphamide. Patients in the this will receive cyclophosphamide 50 mg daily plus letrozole 2.5 mg daily.
  Interventions: Drug: Cyclophosphamide 50mg; Drug: Letrozole 2.5 mg
- Cyclophosphamide plus letrozole for treat-naive patients (Experimental): Patients who haven't received letrozole hormonotherapy will be randomized to receive letrozole plus cyclophosphamide or letrozole alone. Patients in this arm will receive cyclophosphamide 50 mg daily plus letrozole 2.5 mg daily.
  Interventions: Drug: Cyclophosphamide 50mg; Drug: Letrozole 2.5 mg
- letrozole alone (Active Comparator): Patients who haven't received letrozole hormonotherapy will be randomized to receive letrozole plus cyclophosphamide or letrozole alone. Patients in this arm will receive letrozole 2.5 mg daily.
  Interventions: Drug: Letrozole 2.5 mg

INTERVENTIONS:
Drug: Cyclophosphamide 50mg
  Arms: Cyclophosphamide alone; Cyclophosphamide plus letrozole for resistant patients; Cyclophosphamide plus letrozole for treat-naive patients
Drug: Letrozole 2.5 mg
  Arms: Cyclophosphamide plus letrozole for resistant patients; Cyclophosphamide plus letrozole for treat-naive patients; letrozole alone

SUMMARY:
This is a randomized clinical trial to investigate the efficacy of letrozole combined with metronomic oral cyclophosphamide in elderly metastasis breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic breast cancers patients with estrogen receptor positive and/or progesterone receptor positive;
* Elderly women (age ≥ 65years)
* Failure or relapse from standard chemotherapy or unfit for chemotherapy
* Measurable disease per Response Evaluation Criteria in Solid Tumors(RECIST);
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
* Adequate bone marrow, liver and renal function;
* Estimated life expectancy of at least 3 months.

Exclusion Criteria:

* Serious or uncontrolled concurrent medical illness
* Uncontrolled primary and metastatic brain tumor
* History of second primary malignancies
* Having been enrolled in other clinical trials within a month

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2020-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Progression free survival(PFS) of the subjects | up to approximately 2 years
  Time from the randomization date to the start of disease progression or subject death from any cause (progression assessed by investigator using Response Evaluation Criteria in Solid Tumors 1.1for elderly metastatic breast cancer subjects).

SECONDARY OUTCOMES:
Safety of each treatment regimen for the subjects | up to approximately 2 years
  Assessment based on Adverse Events (AEs) , Serious Adverse Events (SAEs), laboratory abnormalities in subjects .
Evaluate the quality of life for the subjects in the each treatment regimen | up to approximately 2 years
  Subjects complete questionnaire in every 8 weeks.
Compare disease control rate for the subjects | up to approximately 2 years
  Complete response (CR), Partial response (PR), and Stable Disease (SD) more than or equal to 8 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Capital Medical Unvierstiy Cancer Center/ Beijing Shijitan Hospital, Beijing, China